CLINICAL TRIAL: NCT01795430
Title: A Pilot Study of Whole-body MRI-guided Intensity Modulated Radiation Therapy Combined With Systemic Chemotherapy Followed by High-Dose Chemotherapy With Busulfan, Melphalan and Topotecan and Stem Cell Rescue in Patients With Poor Risk Ewing's Sarcoma
Brief Title: Whole-Body Radiation Therapy, Systemic Chemotherapy, and High-Dose Chemotherapy Followed By Stem Cell Rescue in Treating Patients With Poor-Risk Ewing Sarcoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled.
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12391; NCI-2013-00439 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Adult Supratentorial Primitive Neuroectodermal Tumor (PNET); Ewing Sarcoma of Bone; Extraosseous Ewing Sarcoma; Metastatic Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Childhood Supratentorial Primitive Neuroectodermal Tumor; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Untreated Childhood Supratentorial Primitive Neuroectodermal Tumor
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive, Peripheral | interventions — Etoposide; Ifosfamide; indolepropanol phosphate; Radiotherapy, Intensity-Modulated; Topotecan; trioctyl phosphine oxide; Busulfan; Melphalan; Peripheral Blood Stem Cell Transplantation; Bone Marrow Transplantation; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (radiation therapy/chemotherapy, stem cell infusion) (Experimental): BLOCK I: Patients receive etoposide IV over 1-2 hours and ifosfamide IV over 1 hour on days 1-5. Patients also undergo WB-MRI-guided intensity-modulated radiation therapy BID, 5 days a week, for approximately 4 weeks. Patients may also undergo 4 fractions of SRT QOD, 3-8 fractions of SBRT QOD, or 10 fractions of 3D RT daily to sites of metastatic disease.
  BLOCK II: Patients receive high-dose chemotherapy comprising topotecan hydrochloride IV continuously over 24 hours on days -8 to -4, busulfan IV over 2 hours every 6 hours on days -8 to -4, and melphalan IV over 30 minutes on days -3 and -2. Patients undergo autologous peripheral blood or bone marrow stem cell infusion on day 0.
  Interventions: Drug: etoposide; Drug: ifosfamide; Radiation: intensity-modulated radiation therapy; Drug: topotecan hydrochloride; Drug: busulfan; Drug: melphalan; Procedure: autologous hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Procedure: autologous bone marrow transplantation

INTERVENTIONS:
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: ifosfamide — Given IV
  Other Names: Cyfos; Holoxan; IFF; IFX; IPP
Radiation: intensity-modulated radiation therapy — Undergo WB-MRI-guided IMRT
  Other Names: IMRT
Drug: topotecan hydrochloride — Given IV
  Other Names: hycamptamine; Hycamtin; SKF S-104864-A; TOPO
Drug: busulfan — Given IV
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon
Drug: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin
Procedure: autologous hematopoietic stem cell transplantation — Undergo autologous peripheral blood stem cell or bone marrow transplant
Procedure: peripheral blood stem cell transplantation — Undergo autologous peripheral blood stem cell transplant
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Procedure: autologous bone marrow transplantation — Undergo autologous bone marrow transplant
  Other Names: ABMT; bone marrow transplantation, autologous; transplantation, autologous bone marrow

SUMMARY:
This pilot clinical trial studies whole-body radiation therapy, systemic chemotherapy, and high-dose chemotherapy followed by stem cell rescue in treating patients with poor-risk Ewing sarcoma. Giving chemotherapy and radiation therapy before a peripheral blood stem cell or bone marrow transplant stops the growth of tumor cells by stopping them from dividing or killing them. After treatment, stem cells are collected from the patient's blood and stored. More chemotherapy is given to prepare the bone marrow for stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and feasibility of whole-body magnetic resonance imaging (WB-MRI)-guided intensity modulated radiation therapy delivered concurrently with systemic chemotherapy to sites of metastatic disease in patients with relapsed, refractory and/or poor risk Ewing sarcoma.

II. To assess the safety and feasibility of a novel consolidation regimen consisting of busulfan, melphalan and topotecan (topotecan hydrochloride) followed by autologous stem cell rescue, to be administered immediately after completion of radiation therapy in patients with relapsed, refractory and/or poor risk Ewing sarcoma.

SECONDARY OBJECTIVES:

I. To characterize the timing of myeloid and platelet engraftment.

II. To estimate the overall and progression free survival probabilities.

III. To estimate the cumulative incidence of relapse/progression and non-relapse related mortality.

IV. To report the overall response rate (overall response rate [ORR]: complete response [CR]+partial response [PR]) and response duration.

V. To descriptively compare the diagnostic imaging results (number and site of bone metastases) of whole-body MR imaging to those obtained by skeletal scintigraphy.

OUTLINE:

BLOCK I: Patients receive etoposide intravenously (IV) over 1-2 hours and ifosfamide IV over 1 hour on days 1-5. Patients also undergo WB-MRI-guided intensity-modulated radiation therapy twice daily (BID), 5 days a week, for approximately 4 weeks. Patients may also undergo 4 fractions of stereotactic radiation therapy (SRT) every other day (QOD), 3-8 fractions of stereotactic body radiation therapy (SBRT) QOD, or 10 fractions of 3-dimensional radiation therapy (3D RT) daily to sites of metastatic disease.

BLOCK II: Patients receive high-dose chemotherapy comprising topotecan hydrochloride IV continuously over 24 hours on days -8 to -4, busulfan IV over 2 hours every 6 hours on days -8 to -4, and melphalan IV over 30 minutes on days -3 and -2. Patients undergo autologous peripheral blood or bone marrow stem cell infusion on day 0.

After the stem cell infusion, patients are followed up for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed Ewing's sarcoma or primitive neuroectodermal tumor (PNET) with bony/soft tissue metastasis who achieved at least partial response (PR) to chemotherapy, surgery or radiotherapy
* Newly diagnosed patients with metastatic disease to the bones: patients with metastatic Ewing's or metastatic PNET who achieved at least partial response (PR) to chemotherapy, surgery or radiotherapy are eligible
* Ewing's sarcoma/PNET histology confirmed by Anatomic Pathology Department; histological confirmation of relapse is highly recommended but not mandatory
* Patients must have documented at least partial response (PR) to previous therapy regimens; previous modalities may include surgery, chemotherapy, or radiation therapy; radiation must not include lung fields; only patients in CR or PR at the primary site will be eligible
* Patients must have metastatic/recurrent disease identified by WB-MRI at the time of study entry; intensity-modulated radiation therapy (IMRT) can be delivered per protocol guidelines to at least one but not more than five primary/metastatic sites
* Patients must have Karnofsky performance status > 60% OR Lansky performance status > 50% for patients younger than 16 years old
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Adequate number of autologous stem cells collected and cryopreserved prior to starting the study treatment
* Creatinine clearance (12 or 24 hour urine collection) or glomerular filtration rate (GFR) > 60 ml/min/1.73 m^2
* Ejection fraction > 50% by echocardiogram or multiple gated acquisition (MUGA)
* Bilirubin < 2 x upper limit of normal
* Serum glutamic oxalo-acetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) < 5 x upper limit of normal
* Platelet count > 50,000/ul
* Absolute granulocyte count >= 750/ul
* Forced expiratory volume in one second (FEV1) > 2 liters adults (older than 16 years)
* Room air arterial oxygen pressure (PaO2) > 70 mm Hg adults (older than 16 years)
* Room air partial pressure of carbon dioxide (PaCO2) < 42 mm Hg adults (older than 16 years)
* Diffusion capacity of carbon monoxide (DLCO) > 50% predicted
* If unable to cooperate with pulmonary function testing due to young age, then pulse oximetry >= 94% children (younger than 16 years)
* Pretreatment tests must have been performed within 4 weeks prior to initiation of protocol treatment
* No other medical and/or psychosocial problems which, in the opinion of the primary physician or principal investigator, would place the patient at unacceptable risk from this regimen
* Greater than 2 week period of recovery from prior modality used to control primary or recurrent site
* All subjects or their legal guardians must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active infection
* Patients may not be receiving any other investigational agents, concurrent biological agents, or chemotherapy
* Patients must not have received prior chemotherapy or radiation within 2 weeks before study enrollment, and those who have not recovered from the adverse events due to agents administered more than 2 weeks earlier are excluded
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated on this study
* Patients with other active malignancies are ineligible for this study
* Patients with prior treatment with myeloablative therapy are excluded
* Karnofsky performance status < 60% or Lansky performance status < 50% for patients younger than 16 years old
* Patients who require irradiation to more than 5 disease sites are excluded
* Subjects who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Ages: 6 Months to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who experience grade 4-5 non-hematologic toxicities assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to day 100 of Block II
  Toxicities will be summarized as type, severity, date of onset, duration, reversibility, and attribution.

SECONDARY OUTCOMES:
Overall response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 5 years
  Objective tumor response for all patients will be summarized, including the number and percent responding.
Progression-free survival (PFS) | Time from stem cell infusion to the first observation of disease progression or death from any cause, whichever occurs first, assessed up to 5 years
  PFS will be estimated using the Kaplan-Meier product-limit method; 95% confidence intervals (CIs) will be calculated using the logit transformation and the Greenwood variance estimate.
Overall survival (OS) | Time from stem cell infusion to death from any cause, assessed up to 5 years
  OS will be estimated using the Kaplan-Meier product-limit method; 95% confidence intervals (CIs) will be calculated using the logit transformation and the Greenwood variance estimate.
Non-relapse mortality (NRM) | Time from stem cell infusion to death event where the cause of death is not attributable to the underlying disease, assessed up to 5 years
  Cumulative relapse incidence will be estimated treating non-relapse related death events as competing risks and, conversely, NRM will be calculated controlling for relapse as a competing risk. Cumulative incidence of NRM and relapse-related mortality will be calculated using the method of Goole et al. Cumulative incidence differences will be assessed by Gray's test.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Pawlowska, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States